CLINICAL TRIAL: NCT05487573
Title: Performance of the Variation in Arterial Lactatemia During a Spontaneous Breathing Trial (SBT) in the Prediction of Extubation Failure
Acronym: PREDILACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00111-42
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-07

CONDITIONS: Extubation Failure
Keywords: Extubation failure; spontaneous breathing trial (SBT); lactatemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extubation failure (EF) is independently associated with excess mortality of critically ill patients. To avoid EF, critically ill patients being weaned from invasive mechanical ventilation (IMV) perform spontaneous breathing trial (SBT), which is the litmus test for determining the ability to breathe without a ventilator.

Thus, the performance of the SBT during weaning from IMV to predict successful extubation is crucial. The investigators hypothesize that patients with EF increase arterial lactate concentration during SBT due to increased work of breathing and hypoxia.

The aim of this study is to evaluate the performance of variation in arterial lactate concentration before and after SBT in predicting successful extubation in critically ill patients.

DETAILED DESCRIPTION:
Extubation failure (EF) is defined as the need for reintubation within 48-72 hour. This complication is independently associated with a seven-fold increased risk of death in critically ill patients.

To avoid EF, critically ill patients being weaned from invasive mechanical ventilation (IMV) perform spontaneous breathing trial (SBT), which is the litmus test for determining the ability to breathe without a ventilator. However, EF occurs in 10 to 20% of patients despite having successful SBT.

Thus, the performance of the SBT during weaning from IMV to predict successful extubation is crucial.

Previous studies of predictive markers of EF have been performed primarily to assess weaning failure from cardiac origin.

The investigators hypothesize that critically ill patients who are going to have EF increase arterial lactate concentration during SBT due to increased work of breathing and hypoxia, regardless of the cause of failure.

The aim of this study is to evaluate the performance of variation in arterial lactate concentration before and after SBT in predicting successful extubation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Intubation and ventilation > 24 hours

Exclusion Criteria:

* Patients under guardianship or curators
* Opposition to participation in the study by the patient or family member
* Patients with tracheotomy
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in intensive care, on invasive mechanical ventilation for more than 24 hours, and performing a spontaneous ventilation trial will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the variation in arterial lactate concentration | 72 hours
  Evaluation of the variation in arterial lactate concentration measured before and after spontaneous ventilation trial in during weaning from invasive mechanical ventilation to predict extubation failure.

SECONDARY OUTCOMES:
Arterial lactate concentration before the spontaneous ventilation trial | 30 minutes
  Measurement of arterial lactate concentration (mmol/L) before the spontaneous ventilation trial.
Arterial lactate concentration after the spontaneous ventilation trial | 30 minutes
  Measurement of arterial lactate concentration (mmol/L) after the spontaneous ventilation trial and before reconnection to mechanical ventilation.
Diagnostic performance of the variation in arterial lactate concentration | 72 hours
  Calculation of the area under the receiver operating characteristic curves (AUROC) for the variation in arterial lactate concentration measured before and after spontaneous ventilation trial.

CONTACTS AND LOCATIONS:
Overall Officials: Alexy Tran Dinh, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat - Claude-Bernard hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided